CLINICAL TRIAL: NCT05952284
Title: Couples Health Aging, Rhythms and Sleep Study (CHARMS Study)
Brief Title: Couples Health Aging, Rhythms and Sleep Study
Acronym: CHARMS
Status: Active, not recruiting | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Kelly Glazer Baron, Associate Professor, PhD, MPH, University of Utah
Other Study IDs: IRB_00158095
Record Dates: First submitted 2023-06-20; First posted 2023-07-19 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Aging; Memory Loss
Keywords: aging; memory; sleep; circadian rhythms
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Alzheimer's disease and related dementias (ADRD), including mild cognitive impairment (MCI), are becoming among the most prevalent causes of disability, death and healthcare costs worldwide. Sleep and circadian rhythm disturbances are common among individuals with MCI as well as their spouses/ partners and may increase risk of the development of ADRD in both patients and partners. This is the first study to systematically investigate sleep as a shared health behavior within couples in which one member has MCI, and the degree to which sleep and circadian disturbances impact both partners health and well-being, including cognitive decline and risk for ADRD.

DETAILED DESCRIPTION:
Individuals with mild cognitive impairment (MCI) demonstrate cognitive decline without major functional impairment but also experience a 7-fold increased risk for developing Alzheimer's disease, a leading cause of poorer quality of life (QOL), premature mortality, and health care expenditures. Sleep and biobehavioral rhythm disturbances (disruptions in 24h oscillations in physiology and behavior, including rest-activity patterns and mealtimes) are more than twice as common among patients with MCI than cognitively intact older adults. Emerging evidence demonstrates a mechanistic role of sleep and biobehavioral rhythm disturbances in cognitive decline and the development and progression of Alzheimer's disease. Importantly, the consequences of sleep and biobehavioral rhythm disruption in MCI extend beyond the patient, also affecting the spouse/partner, as sleep is a "shared" health behavior for most adults. However, sleep and biobehavioral rhythms are typically considered at the level of the individual.

The overall goal of the study is to investigate sleep and biobehavioral rhythms as fundamental dyadic processes that contribute to the health and cognitive functioning of individuals with MCI or mild AD and their partners. The project will evaluate the daily and longitudinal effects of two dyadic processes in sleep:interdependence (partners' sleep patterns influence on each other) and concordance (i.e., the couples' similarity in rest/activity and social rhythms such as meal timing). The protocol involves a 14-day naturalistic study protocol in order to examine the mechanistic associations between sleep and biobehavioral rhythms and proximal indicators of daytime functioning, within a sample of 170 couples in which one partner evidences cognitive impairment (MCI to mild Alzheimer's disease). During the naturalistic study protocol, measures will capture sleep and biobehavioral rhythms via objective (actigraphy) measures of sleep and circadian rest-activity rhythms and daily social rhythms, respectively. Also, measures include daily assessments of mood and relationship quality and an an innovative smartphone cognitive assessment that has been validated to measure cognitive function in daily life. The longitudinal assessment will include comprehensive neuropsychological assessments at baseline and again at two-year follow-up to examine how sleep and biobehavioral rhythm disruptions at baseline predict cognitive decline over 2 years in both partners.

Results of study will advance the understanding of the daily and longitudinal relationships between the individual and couple-level processes in sleep and biobehavioral rhythms that influence the progression of cognitive decline in a population at increased risk for developing Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Married or partnered in a romantic relationship, cohabiting for at least two years
* age >50
* smartphone user
* one partner meets criteria for cognitive impairment without severe impairment in daytime dysfunction according to telephone screening, while other partner must not meet this criteria for impairment.

Exclusion Criteria:

* Unstable or severe medical or psychiatric conditions that would interfere with study participation (including but not limited to current cancer treatment, psychosis, history of major stroke, head injury with loss of consciousness >30 min, other neurologic/systemic illness that may affect cognition, alcohol or other substance abuse)
* current use of antipsychotic or anticonvulsant medications
* inadequate vision, hearing, or dexterity to participate in the assessment
* night shift work >1x per month (defined as beginning work after 9:00 pm or work in the overnight hours [12:00 am-5:00 am])

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be married or cohabiting couples recruited from community locations in the United States who meet the study criteria.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2027-10-02 (Estimated)

PRIMARY OUTCOMES:
Digit symbol: daily score | This study will evaluate day to day change in digit symbol performance over 10 days.
  This is a daily measure of attention and processing speed collected via smartphone. Participants will have 5 minutes to complete the items. In this measure, participants match each symbol presented to a number. The goal of the test is to complete the most items in the time allotted.
Memory: daily score | This study will evaluate day to day change in digit symbol performance over 10 days.
  In this measure, participants will have the opportunity to learn a set of 18 words (30 seconds). These words will be present later in the assessment and participants are asked to recognize whether they are on the list.

SECONDARY OUTCOMES:
Cogntive function: RBANS total score | We will evaluate change from baseline to two years
  We will administer a standardized test battery called the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). This test takes approximately 30 min and measures the main domains of cognitive function, including immediate memory, visuospatial/construction, language, attention, delayed memory and effort

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Data available upon request.